CLINICAL TRIAL: NCT04067895
Title: Multi-center Observational Study on the Use of a Human Bone Graft in Epiphysiodesis
Brief Title: Human Bone Graft in Epiphysiodesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Surgebright Gmbh (Industry)
Responsible Party: Principal Investigator, Catharina Chiari, Univ. Prof. Dr. Catharina Chiari, MSc, Medical University of Vienna
Other Study IDs: EP1
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Leg Length Differences; Primordial Gigantism
Keywords: human bone graft screw; epiphysiodesis; leg length inequality; primordial gigantism
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- human bone graft screw: human bone graft screws will be used during the epiphysiodesis
  Interventions: Procedure: epiphysiodesis

INTERVENTIONS:
Procedure: epiphysiodesis — All patients undergo surgical treatment of leg lengths discrepancies or primordial gigantism. Human bone graft screws will be used to stop the distraction of the growth plate.

SUMMARY:
This observational study is to document the application of human bone graft in the surgical treatment (epiphysiodesis) of leg length discrepancy or primordial gigantism and its subsequent healing process.

ELIGIBILITY:
Inclusion Criteria:

* Planned epiphysiodesis to stop the growing of a bone indicated by leg length discrepancies or primordial gigantism
* Age 10-18 years
* Written consent to participate in the study after previous written and oral education (additional consent for the participation of minors in the study after prior written and oral education by at least one parent)

Exclusion Criteria:

* Insufficient knowledge of the german language
* Foreseeable compliance issues
* Neoplastic diseases, malignant bone tumors, rheumatoid arthritis
* Patients with non-treated pre-existing conditions, which could be the cause of leg length differences
* Active osteomyelitis
* Ulcerations in the area of the skin of the surgical area
* Immunosuppressive drugs that can not be discontinued

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from all participating sites scheduled for an epiphysiodesis with humanm bone graft screws get information about this observational study and have the possibiltiy to participate.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
formation of a bone bridge | 1 year
  based on x-rays or MRI: Is as formation of a bone bridge visible? YES/NO How many millimeters? mm
incidence of surgical revisions | 1 year
  Was a surgical revision done postoperatively? YES/NO
incidence of additional surgery | 1 year
  Was an additional surgery necessary to stop growth? YES/NO; Which one?
incidence of cracking of the screw | 1 year
  based on x-rays or MRI: Is a crack of the screw visible? YES/NO
incidence of a dislocation of the screw | 1 year
  based on x-rays or MRI: Is the screw dislocated? YES/NO
incidence of postoperative inflammatory complications | 1 year
  Is a postoperative inflammatory complication recognizable? YES/NO
cystic brightening around the screw | 1 year
  based on x-rays or MRI: Is a cystic brightening around the screw visible? YES/NO
sclerosing around the screw | 1 year
  based on x-rays or MRI: Is a sclerosis around the screw visible? YES/NO
evaluation of postoperative pain (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = no pain - 100mm = worst imaginable pain). A higher score indicates more pain.

SECONDARY OUTCOMES:
evaluation of swelling | 1 year
  Is a swelling in the surgery area visible? NO/MILD/MODERATE/SEVERE
evaluation of wound healing disorder | 1 year
  Is a disorder of the wound healing recognizable? NO/MILD/MODERATE/SEVERE
evaluation of hematoma | 1 year
  Is a hematoma in the surgery area visible? NO/MILD/MODERATE/SEVERE
patient satisfaction (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = very satisfied - 100mm = not satisfied at all). A higher score indicates less satisfaction.
Knee Outcome Survey - Activities of Daily Living Scale (KOS-ADL) | 1 year
  The KOS ADL score includes 14 questions and is divided in 2 subscales, symptoms (6 items, max. score 30) and functional restrictions (8 items, max. score 40). The scores of the answers range from 0 to 5 points. 0 points mean no impairment of everyday activities, while 5 points represent the greatest possible impairment. All points are summed up.
  From this, the KOS-ADL score is calculated as the proportion of the total response points from the possible maximum score (70) in percent. KOS ADL Score [%] = ( symptoms pts. + functional restrictions pts.)*100/70. The percentage ranges from 0-100%. 0% means no impairment, while 100% represents the greatest possible impairment.
International Knee Documentation Committee Subjective Knee Form (IKDC Score) | 1 year
  The IKDC Score contains 19 questions (7 questions for symptomatology, 10 concerning function, 2 about sport activity). The lowest function level or the highest symptom level receives the score value 1. The highest function level or the lowest symptom level is given the number n according to the number n of possible answers. With the exception of question 10 "Functioning before knee injury", the remaining 18 response points are summed up. This gives the "raw sum". The lowest possible score is 18 and the maximum possible score is 87. The raw sum is converted into a scale of 0 to 100 using the following formula: ((raw score - lowest possible score)/score range)*100. 0 points mean the greatest possible impairment, while 100 points mean complete freedom from symptoms and functioning. The IKDC score can only be calculated if at least 16 of the 18 questions have been answered.
Revised questionnaire to assess Health-Related Quality of Life in children and adolescents (KINDL) | 1 year
  The KINDL is a generic instrument for assessing Health-Related Quality of Life in children and adolescents aged 3 years and older. There are 3 versions available for different age groups: Kiddy-KINDL 4-6 years, Kid-KINDL 7-13 years, Kiddo-KINDL 14-17 years. The questionnaires used in this study (Kid-KINDL and Kiddo-KINDL) provide 24 Likert-scaled items associated with 6 dimensions: physical well-being ,emotional well-being, self-esteem, family, friends, and school. All versions also contain an additional section 'disease' with 6 items. They can be completed in case of illness or hospitalization. The items and sub-scales are calculated according to the KINDL manual and a higher score corresponds to a higher health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Vienna, Vienna, Austria